CLINICAL TRIAL: NCT00258856
Title: Persistence of Bactericidal Antibodies in Children Aged 7 to 15 Years Who Received a Single Dose of Menactra® or Menomune®-A/C/Y/W-135 Five Years Earlier
Brief Title: Persistence of Antibodies in Children Aged 7 to 15 Years Who Previously Received One Dose of Menactra® or Menomune®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA23
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Results first posted 2009-11-25 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Meningitis; Meningococcal Infection
Keywords: Meningitis; Meningococcal infection; Neisseria meningitidis; Menactra®; Menomune®
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Haemophilus influenzae type b-polysaccharide vaccine-diphtheria toxoid conjugate; Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Menactra® Group 1 (Experimental): Participants who had received Menactra® in Study 603-02. They will provide serum sample before vaccination and on Day 3 and Day 7 after booster vaccination.
  Interventions: Biological: Polysaccharide Diphtheria Conjugate Vaccine
- Menactra® Group 2 (Experimental): Participants who had received Menactra® in Study 603-02. They will provide serum sample before vaccination and on Day 5 and Day 14 after booster vaccination.
  Interventions: Biological: Polysaccharide Diphtheria Conjugate Vaccine
- Meningococcal Vaccine-naïve Group 3 (Experimental): Participants who have never received a Meningococcal vaccine in the past. They will provide serum sample before vaccination and on Day 3 and Day 7 after Menactra® vaccination.
  Interventions: Biological: Polysaccharide Diphtheria Conjugate Vaccine
- Meningococcal Vaccine-naïve Group 4 (Experimental): Participants who have never received a Meningococcal vaccine in the past. They will provide serum sample before vaccination and on Day 5 and Day 14 after Menactra® vaccination.
  Interventions: Biological: Polysaccharide Diphtheria Conjugate Vaccine

INTERVENTIONS:
Biological: Polysaccharide Diphtheria Conjugate Vaccine — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Group 1
Biological: Polysaccharide Diphtheria Conjugate Vaccine — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Group 2
Biological: Polysaccharide Diphtheria Conjugate Vaccine — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Meningococcal Vaccine-naïve Group 3
Biological: Polysaccharide Diphtheria Conjugate Vaccine — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Meningococcal Vaccine-naïve Group 4

SUMMARY:
The study is designed to evaluate the persistence of bactericidal antibodies in subjects aged 7 to 15 years (not yet 16 years) who had been vaccinated five years previously in Study 603-02. In addition, the kinetics of the antibody response will be evaluated in a subset of participants who will receive a booster dose of Menactra® vaccine and children in the same age group not previously vaccinated with a meningococcal vaccine or had meningitis disease who will receive a dose of Menactra® vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy, as determined by medical history.
* Subject is between the ages of 7 and 15 years (not yet 16 years).
* For subjects who participated in Study 603-02, subject previously received one dose of Menactra® vaccine or Menomune®-A/C/Y/W-135 vaccine.
* The date of vaccination during Study 603-02 will have occurred 5 years ± 6 months before the collection of the blood sample obtained for Study MTA23.
* A negative urine pregnancy test is required for menstruating female subjects.
* Parent/legal guardian has signed an Institutional Review Board (IRB)-approved informed consent form and subject has signed an IRB-approved assent form.

Exclusion Criteria:

* Subjects who participated in sanofi pasteur Study MTA17 Stage I (a subset of subjects from Study 603-02 who had been recruited for the follow-up challenge study)
* History of documented invasive meningococcal disease
* Received any other meningococcal vaccine
* Received any vaccine in the 28-day period prior to enrollment
* Received antibiotic therapy within the 72 hours prior to collection of a blood sample
* Actively enrolled or scheduled to be enrolled in another clinical study
* Serious chronic disease (i.e., cardiac, renal, neurologic, rheumatologic, metabolic, gastrointestinal, psychiatric, or other organ system)
* Known or suspected impairment of immunologic function
* Acute medical illness with or without fever within 72 hours or an oral temperature ≥ 100.4°F (≥ 38.0°C) at the time of inclusion
* Scheduled to receive any vaccination in the 7-day or 14-day period after enrollment
* Administration of immune globulin, other blood products, or corticosteroid within 8 weeks (56 days) of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting < 7 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment.
* Personal of family history of Guillain-Barres Syndrome
* Suspected or known hypersensitivity to any of the vaccine components
* Unavailable for the entire study period or unable to attend the scheduled visits or to comply with the study procedures
* Any condition which, in the opinion of the investigator, would pose a health risk to the participant.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 234 (Actual)
Dates: Start 2006-01; Primary Completion 2007-03 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (11):
- United States (11):
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Marietta, Georgia
  - Baltimore, Maryland
  - Woburn, Massachusetts
  - Bridgeton, Missouri
  - Rochester, New York
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Salt Lake City, Utah
  - Norfolk, Virginia

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in 18 US clinic sites from 14 January 2006 through 05 June 2006.
Pre-assignment Details: A total of 234 participants that met the inclusion but none of the exclusion criteria were enrolled and vaccinated.
Groups:
- Menactra® Group 1: Participants received Menactra® in Study 603-02.
  Participants provided serum sample before vaccination and on Day 3 and Day 7 after booster vaccination
- Menactra® Group 2: Participants received Menactra® in Study 603-02.
  Participants provided serum sample before vaccination and on Day 5 and Day 14 after booster vaccination
- Meningococcal Vaccine-naïve Group 3: Participants have never received a Meningococcal vaccine in the past. Participants provided serum sample before vaccination and on Day 3 and Day 7 after Menactra® vaccination.
- Meningococcal Vaccine-naïve Group 4: Participants have never received a Meningococcal vaccine in the past. Participants provided serum sample before vaccination and on Day 5 and Day 14 after Menactra® vaccination.
Period: Overall Study
Arm/Group | Menactra® Group 1 | Menactra® Group 2 | Meningococcal Vaccine-naïve Group 3 | Meningococcal Vaccine-naïve Group 4
Started | 59 | 58 | 58 | 59
Completed | 56 | 58 | 56 | 58
Not Completed | 3 | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0
Not completed — Non-compliance | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menactra® Group 1 | Menactra® Group 2 | Meningococcal Vaccine-naïve Group 3 | Meningococcal Vaccine-naïve Group 4 | Total
Number analyzed (Participants) | 59 | 58 | 58 | 59 | 234
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59 | 58 | 58 | 59 | 234
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (2.56) | 10.6 (2.60) | 11.7 (2.27) | 11.9 (2.06) | 11.0 (2.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 25 | 23 | 96
  Male | 33 | 36 | 33 | 36 | 138
Region of Enrollment [Number; unit: participants]
  United States | 59 | 58 | 58 | 59 | 234

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Bactericidal Activity of ≥ 1:8 for the Menactra® Meningococcal Serogroups Pre-vaccination, and at 7 Days or 14 Days Post-booster or Post-primary Dose Vaccination.
Description: Groups 1 and 2 received booster vaccination; Groups 3 and 4 received primary vaccination.
  Serum bactericidal activity for the Menactra® meningococcal serogroups A, C, Y, and W-135 were at pre-vaccination for all Groups, and at 7 days (Groups 1 and 3), and 14 days (Groups 2 and 4) post-vaccination.
Time Frame: 7 or 14 days post-vaccination
Population: Serum bactericidal assay performed using baby rabbit complement (SBA-BR) titers for each of the 4 meningococcal serogroups in the vaccine was evaluated in the per-protocol population.
Measure: Number; unit: Percentage of participants
Arm/Group | Menactra® Group 1 | Menactra® Group 2 | Meningococcal Vaccine-naïve Group 3 | Meningococcal Vaccine-naïve Group 4
Number analyzed (Participants) | 56 | 58 | 56 | 58
Percentage of participants
  Meningococcal serogroup A - PRE | 84 | 89 | 47 | 59
  Meningococcal serogroup A - POST | 100 | 100 | 100 | 100
  Meningococcal serogroup C - PRE | 62 | 58 | 39 | 47
  Meningococcal serogroup C - POST | 100 | 100 | 98 | 96
  Meningococcal serogroup Y - PRE | 96 | 96 | 87 | 98
  Meningococcal serogroup Y - POST | 100 | 100 | 100 | 100
  Meningococcal serogroup W-135 - PRE | 81 | 84 | 31 | 36
  Meningococcal serogroup W-135 - POST | 100 | 100 | 100 | 98

ADVERSE EVENTS:
Time Frame: 28 days post-vaccination
Arm/Group | Menactra® Group 1 | Menactra® Group 2 | Meningococcal Vaccine-naïve Group 3 | Meningococcal Vaccine-naïve Group 4
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58 | 0/58 | 0/59
Other Adverse Events (participants affected / at risk) | 13/58 | 20/58 | 14/58 | 15/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menactra® Group 1 (N=58) | Menactra® Group 2 (N=58) | Meningococcal Vaccine-naïve Group 3 (N=58) | Meningococcal Vaccine-naïve Group 4 (N=59)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 5 (6) | 5 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 1 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 2 (2) | 3 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 4 (4) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 4 (4) | 4 (4)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.